CLINICAL TRIAL: NCT03845985
Title: Piloting "Signs of Safety": A Deaf-Accessible Therapy Toolkit for Alcohol Use Disorder and Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melissa L. Anderson, Associate Professor of Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H00016364; R34AA026929 (NIH)
Record Dates: First submitted 2019-02-01; First posted 2019-02-19 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
Keywords: psychotherapy; trauma; addiction; Deaf
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Wounds and Injuries; Behavior, Addictive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to one of two conditions: (1) Seeking Safety + Signs of Safety toolkit, or (2) assessment-only waitlist control. Randomization will occur within each study site and stratified by gender. The Biostatistician will generate a computerized random number series and place numbers in individual sealed opaque envelopes. The RC will open an envelope to randomly assign a treatment condition to the participant. Both the PI and Co-I/Outcomes Assessor will be blind to study condition. (Note: the Co-I/Outcomes Assessor will remain blind to study condition until the end of the post-treatment assessment, at which point she will administer a client satisfaction measure that will unblind the Co-I to which subjects are in the waitlist control group.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seeking Safety + Signs of Safety toolkit (Experimental): Participants randomized to receive the intervention will be provided 12 one-hour weekly individual treatment sessions with one of four ASL-fluent study clinicians in Massachusetts. Assessments will occur at baseline, week 4, week 8, immediate post-treatment/week 12, and one-month follow-up/week 16.
  Interventions: Behavioral: Seeking Safety + Signs of Safety toolkit
- Assessment-only Waitlist Control (No Intervention): Participants randomized to the waitlist control condition will be offered the opportunity to receive the 12-session Seeking Safety + Signs of Safety toolkit intervention after an approximate 16 week waiting period. This 16 week waiting period is equivalent to the current waitlist to receive psychotherapy services through the PI's outpatient clinic. Assessments will occur at baseline, week 4, week 8, immediate post-treatment/week 12, and one-month follow-up/week 16.

INTERVENTIONS:
Behavioral: Seeking Safety + Signs of Safety toolkit — Seeking Safety is an existing, present-focused, first-stage manualized treatment for trauma and addiction. Session content engages clients in themes relevant to addiction and trauma, and to help them learn a specific skill to target symptoms of both AUD and PTSD (e.g., "Coping with Triggers," "Asking for Help").
  "Signs of Safety" is a culturally and linguistically Deaf-accessible toolkit to be used alongside Seeking Safety. The toolkit includes a therapist guide and population-specific client materials (e.g., visual handouts; ASL teaching stories on digital video). It is designed for Deaf/signing clinicians, as well as non-signing clinicians working with ASL interpreters.
  Arms: Seeking Safety + Signs of Safety toolkit

SUMMARY:
The U.S. Deaf community - more than 500,000 Americans who communicate using American Sign Language (ASL) - experiences nearly triple the rate of lifetime problem drinking and twice the rate of trauma exposure as compared to the general population. Although there are validated treatments for alcohol use disorder (AUD) and post-traumatic stress disorder (PTSD) in hearing populations, there are no evidence-based treatments for any behavioral health condition that have been validated for use with Deaf clients. To address these barriers, the study team has developed "Signs of Safety", a Deaf-accessible therapy toolkit for treating AUD and PTSD. The study team's ongoing aims are to conduct a two-arm pilot RCT of "Signs of Safety" and to collect data on feasibility, preliminary clinical outcomes, and potential mediators and moderators of outcome.

DETAILED DESCRIPTION:
The U.S. Deaf community - 500,000+ Americans who communicate using American Sign Language (ASL) - experiences nearly triple the rate of lifetime problem drinking compared to the general population and twice the rate of trauma exposure. Although there are validated treatments for comorbid alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) in hearing populations, there are no evidence-based treatments to treat any behavioral health condition with Deaf clients. Current treatments fail to meet Deaf clients' unique linguistic and cultural needs. Deaf people's median English reading level falls at the fourth grade, and many have low health literacy due to reduced incidental learning (e.g., inability to communicate with hearing parents, overhear family conversations, or understand spoken health information on TV/radio/public service announcements). Written treatment materials, therefore, require plain text revisions, ASL translations, or ASL narrative storytelling. Equally important are materials that incorporate Deaf values and social norms, increasing clinicians' cultural competence and enhancing client engagement.

To address these barriers, the Principal Investigator conducted a pilot study to develop a prototype of "Signs of Safety": a Deaf-accessible toolkit to be used alongside a widely-disseminated protocol for addiction/PTSD - Seeking Safety. Seeking Safety has demonstrated efficacy for reduction of AUD and PTSD symptoms in hearing populations. Among available evidence-based protocols, "Seeking Safety" is the optimal choice to adapt for Deaf clients - its focus on simple coping skills that simultaneously target AUD and PTSD (or either alone) is an ideal match for Deaf people's language and learning deficits, which prohibit use of verbal problem-solving and cognitive processing strategies that other psychotherapies require. Yet, Seeking Safety's client materials rely on written English and are not well understood by Deaf clients. As such, the "Signs of Safety" toolkit includes a therapist guide and population-specific client materials (e.g., visual handouts; ASL teaching stories on digital video). It is designed for Deaf/signing clinicians, as well as non-signing clinicians working with ASL interpreters.

Data from the Principal Investigator's "Signs of Safety" single-arm pilot study (n = 13) show significant reductions in alcohol use frequency and PTSD severity from baseline to immediate post-treatment follow-up. Participants also reported high levels of satisfaction with the model, and provided detailed feedback about how to further improve "Signs of Safety" for a professional-quality, second iteration. The proposed study builds upon the Principal Investigator's pilot work by generating a final, professional iteration of Signs of Safety to be used in future efficacy work. Based on pilot results, the study team created a second iteration of the "Signs of Safety" toolkit, including re-filming ASL teaching stories, re-designing visual handouts, and revising the therapist companion guide. The study team will then develop a training program for "Signs of Safety" and certify four study clinicians.

The study team proposes to conduct a two-arm pilot RCT of "Signs of Safety". The study team aims to enroll 60 Deaf adults with past-month PTSD and past-month alcohol consumption to participate in 12 weekly individual treatment sessions. The pilot RCT will compare the 12-session protocol of Seeking Safety + "Signs of Safety" toolkit with an assessment-only waitlist control. Across conditions, assessment will occur at baseline, week 4, week 8, immediate post-treatment/week 12, and one-month follow-up/week 16. The study team will analyze key aspects of feasibility for both study arms (e.g., recruitment, retention, assessment process). Primary clinical outcomes at immediate post-treatment and one-month follow-up are past 30-day alcohol use frequency/quantity and past 30-day PTSD severity. Exploratory analyses will be conducted to examine potential moderators and mediators of change (e.g., motivation for treatment, provider cultural competency, coping skills, self-compassion, understanding of health information) leading to positive outcome. Results from this study will produce feasibility and preliminary efficacy data to support for a full-scale RCT to evaluate "Signs of Safety", and a community-engaged model for conducting RCTs with Deaf participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as a Deaf ASL user
* Age 18 or older
* Past-month alcohol consumption, as measured by the Alcohol Use Disorder Identification Test
* Subthreshold or full PTSD on the PTSD Checklist for DSM-5 (past-month referent time period; "subthreshold" = endorsement of at least two B-E criteria at a severity of "moderate" or higher)
* Ability to attend weekly study sessions at one of three study locations (Eastern, Central, or Western MA)
* Ability to access a videophone (the standard telecommunication device for the Deaf community)

Exclusion Criteria:

* Participation in concurrent therapies (Note: Participants in both study conditions will be asked to refrain from concurrent formal psychotherapy; however, aligning with the Seeking Safety model, AA/NA/DRA attendance will be encouraged and attendance will be tracked as a potential outcome mediator).
* Members of the following special populations: Adults unable to consent; Individuals younger than 18; Prisoners; Pregnant women (Note: We will not knowingly include pregnant women as participants; however, we will not assess participants' pregnancy status.)

Exclusion criteria are intentionally minimal to recruit a diverse sample. Other behavioral health comorbidities (e.g., mood/anxiety disorders, substance use disorders other than AUD) will not be excluded, given high rates of comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Anderson, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after deidentification that underlie the reported results (text, tables, figures, and appendices) will be available beginning 9 months and ending 36 months following article publication. Investigators whose proposed use of the data has been approved by an independent review committee may use the data for individual participant data meta-analysis. Proposals may be submitted up to 36 months follow article publication. Please contact the Principal Investigator for information regarding submitting proposals and accessing data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee may use the data for individual participant data meta-analysis.

REFERENCES:
- [Background] Heffernan K. Seeking Safety: A Treatment Manual for PTSD and Substance Abuse. Psychother Res. 2003 Mar;13(1):125-6. doi: 10.1080/713869629. No abstract available. PMID 22475169

RESULTS

PARTICIPANT FLOW:
Groups:
- Seeking Safety + Signs of Safety Toolkit: Participants randomized to receive the intervention will be provided 12 one-hour weekly individual treatment sessions with one of four ASL-fluent study clinicians in Massachusetts. Assessments will occur at baseline, week 4, week 8, immediate post-treatment/week 12, and one-month follow-up/week 16.
  Seeking Safety + Signs of Safety toolkit: Seeking Safety is an existing, present-focused, first-stage manualized treatment for trauma and addiction. Session content engages clients in themes relevant to addiction and trauma, and to help them learn a specific skill to target symptoms of both AUD and PTSD (e.g., "Coping with Triggers," "Asking for Help").
  "Signs of Safety" is a culturally and linguistically Deaf-accessible toolkit to be used alongside Seeking Safety. The toolkit includes a therapist guide and population-specific client materials (e.g., visual handouts; ASL teaching stories on digital video). It is designed for Deaf/signing clinicians, as well as non-signing clinicians working with ASL interpreters.
Period: Overall Study
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Started | 9 | 7
Completed | 2 | 5
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.67 (12.43) | 42.71 (12.16) | 43.81 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
% Drinking Days per Month [Mean (Standard Deviation); unit: percent drinking days per month] — (Number of days per month with 1+ drink) divided by 30 days x 100
  percent drinking days per month | 40.37 (47.74) | 49.52 (46.60) | 44.38 (45.89)
% Binge Drinking Days per Month [Mean (Standard Deviation); unit: percent binge drinking days per month] — (Number of days per month with 5+ drinks for men or 4+ drinks for women) divided by 30 x 100
  percent binge drinking days per month | 16.30 (34.98) | 1.43 (2.62) | 9.79 (26.71)
Total # of Drinks per Month [Mean (Standard Deviation); unit: drinks per month] | 57.89 (89.05) | 42.80 (49.14) | 51.29 (72.49)
Past 30-Day PTSD Severity Score [Mean (Standard Deviation); unit: units on a scale] — Total Score on the PCL-5 divided by 20 items. Minimum score = 0; Maximum score = 4. Higher values represent more severe symptoms of PTSD.
  units on a scale | 1.61 (0.76) | 2.29 (0.68) | 1.91 (0.78)
Brief Comprehensive Effects of Alcohol Score [Mean (Standard Deviation); unit: units on a scale] — All four subscales: Min. = 1, Max. = 4.
  Risk and Aggression/Liquid Courage/Sociability Subscale: Higher values indicate greater outcome expectancies of drinking alcohol on risk-taking, aggression, courage, and sociability.
  Self-Perception/Cognitive and Behavioral Impairment Subscale: Higher values indicate greater outcome expectancies on distorted self-perception and impaired behavior.
  Sexuality Subscale: Higher values indicate greater outcome expectancies on sexual behavior.
  Tension Reduction Subscale: Higher values indicate greater outcome expectancies on tension reduction.
  units on a scale
    Risk and Aggression/Liquid Courage/Sociability Subscale Score | 2.32 (0.99) | 2.67 (0.51) | 2.49 (0.80)
    Self-Perception/Cognitive and Behavioral Impairment Subscale | 1.92 (0.82) | 2.68 (0.81) | 2.25 (0.88)
    Sexuality Subscale | 2.31 (1.44) | 1.57 (0.61) | 1.97 (1.16)
    Tension Reduction | 3.22 (0.67) | 2.93 (0.96) | 3.09 (0.80)
Penn Alcohol Craving Scale Score [Mean (Standard Deviation); unit: units on a scale] — Total score = sum of all 5 items.
  Minimum = 0; Maximum = 30.
  Higher values indicate higher severity of alcohol craving.
  units on a scale | 9.22 (7.85) | 15.43 (3.36) | 11.94 (6.89)
Trauma Symptom Checklist 40 Total Severity Score [Mean (Standard Deviation); unit: units on a scale] — Sum of all items divided by 40 items.
  Minimum = 0; Maximum = 3.
  Higher values indicate more severe trauma symptoms.
  units on a scale | 0.81 (0.34) | 1.47 (0.46) | 1.10 (0.51)
BASIS-24 Total Severity Score [Mean (Standard Deviation); unit: units on a scale] — Sum of all items divided by 24 items.
  Minimum = 0; Maximum = 4.
  Higher values indicate worsening behavior or more severe behavioral health symptoms.
  units on a scale | 1.25 (0.44) | 1.60 (0.44) | 1.40 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Percent Drinking Days Per Month at Immediate Post-Treatment
Description: Change from baseline percent drinking days per month (i.e., days with 1+ drink) at immediate post-intervention or 12 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to immediate post-intervention at 12 weeks
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: percent drinking days per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
percent drinking days per month | -20.00 (29.06) | -11.11 (67.68)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .838, t-test, 2 sided — Analysis was significantly underpowered

2. Primary Outcome: Change From Baseline Percent Drinking Days Per Month at One-month Follow-up
Description: Change from baseline percent drinking days per month (i.e., days with 1+ drink) at one-month follow-up or 16 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to one-month follow-up at 16 weeks
Population: Analysis includes only those participants who completed the one-month follow-up/16 week assessment.
Measure: Mean (Standard Deviation); unit: percent drinking days per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 2 | 5
percent drinking days per month | -26.67 (37.71) | -13.33 (27.99)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .620, t-test, 2 sided — Analysis was significantly underpowered

3. Primary Outcome: Change From Baseline Percent Binge Drinking Days Per Month at Immediate Post-Treatment
Description: Change from baseline percent binge drinking days per month (i.e., days with 5+ drinks for men, 4+ for women) at immediate post-intervention or 12 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to immediate post-intervention at 12 weeks
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: percent binge drinking days per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
percent binge drinking days per month | 17.78 (74.93) | -0.56 (1.36)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .713, t-test, 2 sided — Analysis was significantly underpowered

4. Primary Outcome: Change From Baseline Percent Binge Drinking Days Per Month at One-month Follow-up
Description: Change from baseline percent binge drinking days per month (i.e., days with 5+ drinks for men, 4+ for women) at one-month follow-up or 16 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to one-month follow-up at 16 weeks
Population: Analysis includes only those participants who completed the one-month follow-up/16 week assessment.
Measure: Mean (Standard Deviation); unit: percent binge drinking days per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 2 | 5
percent binge drinking days per month | -23.33 (33.00) | -0.67 (1.49)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .509, t-test, 2 sided — Analysis was significantly underpowered

5. Primary Outcome: Change From Baseline Number of Drinks Per Month at Immediate Post-Treatment
Description: Change from baseline number of drinks per month at immediate post-treatment or 12 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to immediate post-intervention at 12 weeks
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Error); unit: drinks per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
drinks per month | 122.67 (272.56) | -9.17 (40.12)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .491, t-test, 2 sided — Analysis was significantly underpowered

6. Primary Outcome: Change From Baseline Number of Drinks Per Month at One-month Follow-up
Description: Change from baseline number of drinks per month at one-month follow-up or 16 weeks as assessed by Alcohol Timeline Followback
Time Frame: Change from baseline to one-month follow-up at 16 weeks
Population: Analysis includes only those participants who completed the one-month follow-up/16 week assessment.
Measure: Mean (Standard Deviation); unit: drinks per month
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 2 | 5
drinks per month | -33.50 (47.38) | -22.90 (28.04)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .715, t-test, 2 sided — Analysis was significantly underpowered

7. Primary Outcome: Change From Baseline Past 30-day PTSD Severity to Immediate Post-Treatment as Assessed by PCL-5
Description: Total Score on the PCL-5 divided by 20 items. Minimum score = 0; Maximum score = 4. Higher values represent more severe symptoms of PTSD.
Time Frame: Change from baseline to immediate post-intervention at 12 weeks
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
units on a scale | -0.30 (0.05) | -0.53 (0.86)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .665, t-test, 2 sided — Analysis was significantly underpowered

8. Primary Outcome: Change From Baseline Past 30-day PTSD Severity at One-month Follow-up as Assessed by PCL-5
Description: as for outcome 7
Time Frame: Change from baseline to one-month follow-up at 16 weeks
Population: Analysis includes only those participants who completed the one-month follow-up/16 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 1 | 5
units on a scale | -0.40 (NA) — Only 1 participant analyzed in this arm for this outcome. | -0.22 (0.98)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .875, t-test, 2 sided — Analysis was significantly underpowered

9. Secondary Outcome: The Brief Comprehensive Effects of Alcohol Questionnaire (B-CEOA)
Description: All four subscales: Min. = 1, Max. = 4.
  Risk and Aggression/Liquid Courage/Sociability Subscale: Higher values indicate greater outcome expectancies of drinking alcohol on risk-taking, aggression, courage, and sociability.
  Self-Perception/Cognitive and Behavioral Impairment Subscale: Higher values indicate greater outcome expectancies on distorted self-perception and impaired behavior.
  Sexuality Subscale: Higher values indicate greater outcome expectancies on sexual behavior.
  Tension Reduction Subscale: Higher values indicate greater outcome expectancies on tension reduction.
Time Frame: Baseline/Pre-intervention, Week 4, Week 8, Week 12/Post-intervention, and Week 16/One-month Follow-up
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
units on a scale
  Risk and Aggression/Liquid Courage/Sociability Subscale | 0.38 (1.19) | 0.05 (0.73)
  Self-Perception/Cognitive and Behavioral Impairment Subscale | -0.33 (0.38) | 0.00 (1.18)
  Sexuality Subscale | 0.00 (0.00) | 0.00 (0.95)
  Tension Reduction Subscale | 1.83 (0.58) | -0.17 (0.82)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Comparison of the Risk and Aggression/Liquid Courage/Sociability Subscale; Test type: Superiority; p = .610, t-test, 2 sided — Analysis was significantly underpowered
Statistical Analysis 2: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Comparison of the Self-Perception/Cognitive and Behavioral Impairment Subscale; Test type: Superiority; p = .658, t-test, 2 sided — Analysis was significantly underpowered
Statistical Analysis 3: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Comparison of the Sexuality Subscale; Test type: Superiority; p = 1.000, t-test, 2 sided — Analysis was significantly underpowered
Statistical Analysis 4: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Comparison of the Tension Reduction Subscale; Test type: Superiority; p = .007, t-test, 2 sided — Analysis was significantly underpowered

10. Secondary Outcome: Penn Alcohol Craving Scale (PACS)
Description: Total score = sum of all 5 items.
  Minimum = 0; Maximum = 30.
  Higher values indicate higher severity of alcohol craving.
Time Frame: Baseline/Pre-intervention, Week 4, Week 8, Week 12/Post-intervention, and Week 16/One-month Follow-up
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
score on a scale | 1.33 (14.05) | -4.83 (7.62)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .407, t-test, 2 sided — Analysis was significantly underpowered

11. Secondary Outcome: Trauma Symptom Checklist - 40 (TSC-40)
Description: Sum of all items divided by 40 items.
  Minimum = 0; Maximum = 3.
  Higher values indicate more severe trauma symptoms.
Time Frame: Baseline/Pre-Intervention, Week 12/Post-Intervention, Week 16/One-month Follow-up
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 3 | 6
units on a scale | -0.22 (0.31) | -0.15 (0.83)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .893, t-test, 2 sided — Analysis was significantly underpowered

12. Secondary Outcome: Behavior and Symptom Identification Scale - 24 (BASIS-24)
Description: Sum of all items divided by 24 items. Minimum = 0; Maximum = 4. Higher values indicate worsening behavior or more severe behavioral health symptoms.
Time Frame: Baseline/Pre-Intervention, Week 12/Post-Intervention, Week 16/One-month Follow-up
Population: Analysis includes only those participants who completed the immediate post-intervention/12 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
Number analyzed (Participants) | 2 | 6
units on a scale | -0.16 (0.65) | .06 (0.22)
Statistical Analysis 1: Comparison: Seeking Safety + Signs of Safety Toolkit vs Assessment-only Waitlist Control; Test type: Superiority; p = .709, t-test, 2 sided — Analysis was significantly underpowered

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Seeking Safety + Signs of Safety Toolkit | Assessment-only Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

LIMITATIONS AND CAVEATS:
This trial began recruiting in mid-2019. Just as enrollment ramped up, our trial was disrupted by the onset of the COVID-19 pandemic. We paused the study to overhaul our in-person research methods and learn how to implement a virtual clinical trial - an acceleration of the inevitable development needed to scale to a national level. Due to these disruptions, our sample size was small and resulting analyses were significantly underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03845985/Prot_SAP_001.pdf